CLINICAL TRIAL: NCT07113587
Title: Pharmacokinetics of Intraperitoneal and Intravenous Meropenem, Ampicillin, Aztreonam and Ciprofloxacin in Automated Peritoneal Dialysis Patients Without Peritonitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karl Landsteiner Insitute for Nephrology and Haemato-Oncology (Network)
Collaborators: Karl Landsteiner University of Health Sciences (Other); University of Vienna (Other); Medical University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS4-EK-2/301-2013; 2013-004985-32 (EudraCT Number)
Record Dates: First submitted 2025-07-09; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Peritoneal Dialysis-associated Peritonitis; Peritoneal Dialysis (PD); Pharmacokinetics; Intravenous Administration; Intravenous; Meropenem; Intraperitoneal; Ampicillin; Aztreonam; Ciprofloxacin; Minimum Inhibitory Concentration (MIC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ampicillin in APD patients without peritonitis (Experimental)
  Interventions: Drug: Application of intraperitoneal and intravenous ampicillin in automated peritoneal dialysis patients without peritonitis
- meropenem in APD patients without peritonitis (Experimental)
  Interventions: Drug: Application of intraperitoneal and intravenous meropenem in in automated peritoneal dialysis patients without peritonitis
- ciprofloxacin in APD patients without peritonitis (Experimental)
  Interventions: Drug: Application of intraperitoneal and intravenous ciprofloxacin in automated peritoneal dialysis patients without peritonitis
- aztreonam in APD patients without peritonitis (Experimental)
  Interventions: Drug: Application of intraperitoneal and intravenous aztreonam in automated peritoneal dialysis patients without peritonitis

INTERVENTIONS:
Drug: Application of intraperitoneal and intravenous meropenem in in automated peritoneal dialysis patients without peritonitis
  Arms: meropenem in APD patients without peritonitis
Drug: Application of intraperitoneal and intravenous ampicillin in automated peritoneal dialysis patients without peritonitis
  Arms: ampicillin in APD patients without peritonitis
Drug: Application of intraperitoneal and intravenous aztreonam in automated peritoneal dialysis patients without peritonitis
  Arms: aztreonam in APD patients without peritonitis
Drug: Application of intraperitoneal and intravenous ciprofloxacin in automated peritoneal dialysis patients without peritonitis
  Arms: ciprofloxacin in APD patients without peritonitis

SUMMARY:
This study aims to investigate the pharmacokinetics (PK) and pharmacodynamic (PD) profiles of four commonly used antibiotics - meropenem, ampicillin, aztreonam, and ciprofloxacin - administered via intravenous (i.v.) and intraperitoneal (i.p.) routes in patients undergoing automated peritoneal dialysis (APD) without peritonitis. Existing dosing regimens for APD patients are often extrapolated from continuous ambulatory peritoneal dialysis (CAPD) data, despite notable differences in dialysis dynamics, solute clearance, and drug disposition between the two modalities. This discrepancy may result in subtherapeutic exposure or overtreatment, leading to poor clinical outcomes or drug toxicity.

Automated peritoneal dialysis is characterized by multiple, frequent short cycles of dialysate exchange during the night, along with a prolonged daytime dwell using icodextrin-based solutions. These unique features influence both the systemic absorption and elimination of intraperitoneally administered antibiotics. The pharmacokinetics of these antibiotics in APD patients, particularly with regard to intermittent i.p. dosing, remains insufficiently studied.

This single-center, open-label, randomized crossover study will evaluate plasma, dialysate, and urine concentrations of each antibiotic after both i.v. and i.p. administration in 24 adult patients (6 per drug group) receiving APD. Each subject will receive a single dose of one antibiotic (either 0.5g meropenem, 2g ampicillin, 1g aztreonam, or 400mg ciprofloxacin) via both routes, separated by a one-week washout period. Intraperitoneal administration will occur at the end of the cycler session, allowing the drug to dwell in 1.5L of icodextrin solution during the long daytime exchange.

Serial samples of plasma, peritoneal dialysate, and urine will be collected over a 24-hour period following each drug administration. High-performance liquid chromatography (HPLC) will be used to measure drug concentrations. Pharmacokinetic parameters to be calculated include area under the concentration-time curve (AUC), maximum concentration (Cmax), half-life (t½), and time to maximum concentration (Tmax). Secondary PK/PD indices such as time above the minimum inhibitory concentration (T>MIC) and AUC/MIC ratios will also be assessed to estimate the potential efficacy at the infection site.

The study drugs have well-characterized safety profiles and have been previously used via both i.v. and i.p. routes in CAPD and clinical practice. The study protocol includes safety monitoring, including assessment of adverse events, vital signs, hematology, and clinical chemistry parameters. Risks to subjects are considered minimal, primarily related to venous catheterization and single-dose drug administration. Participants are not expected to receive direct therapeutic benefit but will contribute to the optimization of antimicrobial therapy in APD patients with infections such as peritonitis and pneumonia.

This research addresses a critical gap in evidence-based dosing of antimicrobials in the APD population. Results from this study may inform future clinical guidelines and support rational selection and dosing of antibiotics in peritoneal dialysis-associated infections. It also offers insight into the feasibility of intermittent intraperitoneal therapy in APD patients and the systemic exposure achieved through this route. The study is conducted in accordance with Good Clinical Practice (GCP), the Declaration of Helsinki, and Austrian regulatory and ethical requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 on APD using icodextrin.
* Informed consent provided.
* No recent infections or antibiotic use.

Exclusion Criteria

* Active systemic infection or recent peritonitis.
* Severe liver disease, pregnancy, allergy to study drugs.
* Hemoglobin <9 g/dL; BMI <19 or >35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
AUC (Area Under Curve) | 24 hours
Cmax (maximum concentration) | 24 hours
t½ (half-life) | 24 hours
tmax (time to Cmax) | 24 hours

SECONDARY OUTCOMES:
T>MIC (time above minimum inhibitory concentration) | 24 hours
AUC₀-₂₄/MIC ratio | 24 hours
Compartmental AUC/Cmax ratios | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wiesholzer, MD, Principal Investigator — UK St. Pölten - Deparment of Internal Medicine 1, Nephrology
Locations (1):
- UK St. Pölten, Sankt Pölten, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Hextall A, Andrews JM, Donovan IA, Wise R. Intraperitoneal penetration of meropenem. J Antimicrob Chemother. 1991 Aug;28(2):314-6. doi: 10.1093/jac/28.2.314. No abstract available. PMID 1778863
- [Background] Manley HJ, Bailie GR. Treatment of peritonitis in APD: pharmacokinetic principles. Semin Dial. 2002 Nov-Dec;15(6):418-21. doi: 10.1046/j.1525-139x.2002.00103.x. PMID 12437537
- [Background] Van Ende C, Tintillier M, Cuvelier C, Migali G, Pochet JM. Intraperitoneal meropenem administration: a possible alternative to the intravenous route. Perit Dial Int. 2010 Mar-Apr;30(2):250-1. doi: 10.3747/pdi.2009.00052. No abstract available. PMID 20200373
- [Background] Warady BA, Bakkaloglu S, Newland J, Cantwell M, Verrina E, Neu A, Chadha V, Yap HK, Schaefer F. Consensus guidelines for the prevention and treatment of catheter-related infections and peritonitis in pediatric patients receiving peritoneal dialysis: 2012 update. Perit Dial Int. 2012 Jun;32 Suppl 2(Suppl 2):S32-86. doi: 10.3747/pdi.2011.00091. No abstract available. PMID 22851742
- [Background] Li PK, Szeto CC, Piraino B, Bernardini J, Figueiredo AE, Gupta A, Johnson DW, Kuijper EJ, Lye WC, Salzer W, Schaefer F, Struijk DG; International Society for Peritoneal Dialysis. Peritoneal dialysis-related infections recommendations: 2010 update. Perit Dial Int. 2010 Jul-Aug;30(4):393-423. doi: 10.3747/pdi.2010.00049. No abstract available. PMID 20628102
- [Background] Salzer W. Antimicrobial-resistant gram-positive bacteria in PD peritonitis and the newer antibiotics used to treat them. Perit Dial Int. 2005 Jul-Aug;25(4):313-9. PMID 16022084